CLINICAL TRIAL: NCT03675152
Title: Treatment of Spondylolysis With Soft Spinal Brace vs. Boston Brace in Pediatric Patients. A Clinical Trial
Brief Title: Treatment of Spondylolysisin Pediatric Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: Satakunta Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T45/2016
Record Dates: First submitted 2018-08-21; First posted 2018-09-18 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Low Back Pain; Stress Fracture
Keywords: spondylolysis; pediatric
MeSH Terms: conditions — Low Back Pain; Fractures, Stress; Spondylolysis

STUDY DESIGN:
Intervention Model Description: patients are in two groups treated with soft spinal brace or with thoracolumbar orthosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soft spinal brace (Experimental): Soft spinal brace used 23 hours a day for 4 months.
  Interventions: Other: Soft spinal brace; Other: Excersice restriction
- thoracolumbar orthosis (Active Comparator): Thoracolumbar orthosis used 23 hours a day for 4 months.
  Interventions: Other: thoracolumbar orthosis; Other: Excersice restriction

INTERVENTIONS:
Other: Soft spinal brace — Soft thoracolumbar brace worn 23 hours a day.
  Arms: Soft spinal brace
Other: thoracolumbar orthosis — Hard thoracolumbar orthosis done individually molded, Worn 23 hours a day.
  Arms: thoracolumbar orthosis
Other: Excersice restriction — Patients are only allowed to do isometrical excersices adviced by a physiotherapist.

SUMMARY:
A clinical trial comparing healing of unilateral or bilateral spondylolysis in children treated with a Boston thoracolumbar orthosis (brace) or with a soft spinal brace (Porostrap lumbar support) for four months. Inclusion criteria will be a child or adolescent aged between 8 and 20 years with an early uni- or bilateral defect (fracture line) in the pars interarticularis in the CT-scan with no signs of bony sclerosis. Additionally, bone marrow edema has to be confirmed in MR images (T2 sagittal) as a sign of an early lesion. Exclusion criteria will be spondylolisthesis on standing spinal radiograph, systemic skeletal disorder or lack of interest. Patient's preference defines the treatment method. Minimum follow-up time will be 2 years for all patients. According to statistical power analysis a total of 60 patients will be needed to provide evidence for the effectiveness or no effectiveness of rigid thoracolumbar orthosis on the natural history of early spondylolysis. Measured outcome parameters are 1) Bony healing on CT-scan, 2) SRS-24-score at the beginning of the treatment and during the 2-year follow-up, 3) Back and lower extremity pain at the beginning of the treatment and during the 2-year follow-up (Pain drawing including VAS-score in children under 16 years old, Oswestry disability index including VAS-score in patients over 16 years old), 4) Thoracolumbar radiographs at 2-year follow-up: Evidence of spondylolisthesis, 5) Trunk strength and spinal mobility at follow-up visits.

As part of this study, the investigators will also evaluate patients with spondylolysis treated in their hospitals before this clinical trial begun. In this retrospective study they will evaluate all patients between 8 and 20 years of age with spondylolysis, which have been treated with thoracolumbar orthosis after year 2009 and are not participating in to prospective study. Main focus will be in bony healing in CT-scans after brace treatment.

DETAILED DESCRIPTION:
A clinical trial comparing effectiveness of a soft spinal brace and a rigid thoracolumbar orthosis will be performed. Patients will choose the treatment method (patient preference). One option is to be treated, as what is known as a golden standard, with a hard thoracolumbar brace (Boston brace) worn daily for four months. The other option is to be treated with a soft spinal brace for four months. The soft brace we use in this study is DJO Global's Porostrap lumbar support. Both groups cease from sporting activities and get identical physiotherapy, where the aim is to strengthen abdominal and back muscles. After four month brace treatment we will have a control appointment where a CT-scan is taken to detect the bony healing of the pars interarticularis. Other follow-up appointments will be at 12 months and 24 months. Subjective healing is measured each time with SRS-24-score and Oswestry disability Index or pain drawing. During the last appointment, approximately 2 years after beginning of the study, a standing lateral thoracolumbar radiograph is taken to detect if the patient has developed spondylolisthesis. Trunk strength and spinal mobility is measured at follow-up visits (4 months, 12months, and 24months).

SRS-24 questionnaire is a translated and modified version of the Scoliosis Research Society-22 questionnaire. The two first questions measure the intensity of the pain (1 meaning no pain and 9 referring to the worst pain imagined). The remaining 22 questions have five alternatives from 1 (the worst option) to 5 (the best option) and they intend to measure the health-related quality of life. It has been well validated and proved reliable in investigating children with scoliosis quality of life (18).

Oswestry disability Index (ODI) is an index used to evaluate patients' back and lower extremity pain translated in Finnish or Swedish (19). It consists of ten questions and VAS-score. One question is about sexual life and that's why this questionnaire is used only for patients over 16 years old. Patients under 16 years old are asked to fill a pain drawing. This also includes VAS-score.

Visual analogue score (VAS) is a numeric pain distress scale from 0 to 10, where zero refers to "no pain" and ten to " unbearable pain". Patient draws his/her pain in a line from 0 to 10. During each appointment a patient is asked to describe their back pain and/or lower extremity pain in this scale as it is included in both pain drawing and ODI.

Trunk strength and spinal mobility tests are used to evaluate the effect of the use of the brace to the muscles and movement of the trunk. The centimeters with a tape measure from the fingertips on the thigh in side-bend are measured and we grade it abnormal, if the measurement is over 2 standard deviations under the mean of the Finnish reference values (20). Non-dynamometric trunk performance is measured with repetitive sit-up, arch-up and squatting tests. The result is graded from 1 (poor) to 5 (excellent). 1 refers to 1 standard deviation or more below the mean of the normal Finnish population values and 5 to 1 standard deviation or more above this mean (21).

In MRI, from the T2 spin-echo weighted images disc degeneration is graded based on Pfirrmann classification. Grade I refers to normal disc and grade V to most advanced disc degeneration. (22).

Computed tomography (CT) is widely used to diagnose spondylolysis and to detect healing of it. It shows bony healing and nonunion (12). A standing lateral thoracolumbar radiograph is taken at last follow-up visit to determine spondylolisthesis. This is understood as an indirect sign of failure of the treatment of the spondylolysis.

ELIGIBILITY:
Inclusion Criteria:

* Early uni- or bilateral defect in pars interarticularis in the CT-scan
* No signs of bony sclerosis on CT
* No signs of spondylolisthesis on standing lumbar radiographs
* Bone marrow edema in lumbar spinal MR images
* Age between 8 and 20 years
* Written informed consent

Exclusion Criteria:

* Spondylolisthesis
* Systemic skeletal disorder (Osteogenesis imperfecta, skeletal dysplasia)
* Lack of interest

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06-12 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Healing of spondylolysis in computed tomography | 4 months
  Bony healing on 4 month CT-scan measured in three categories: healed, healing in process, not healed.

SECONDARY OUTCOMES:
developement of spondylolisthesis | 2 years
  Lumbar spondylolisthesis at 2-year follow-up
Pain measurement 1: Oswestry disability index | Baseline, 4 months, 12months and 24 months
  Oswestry disability index(patients over 16 years old) 0, 4, 12, 24 months. The self-completed questionnaire contains 10 questions with 6 different answer options. Each question is scored on a scale 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Pain measurement 2 | Baseline, 4 months, 12months and 24 months
  Pain drawing (patients under 16 years old) 0, 4, 12, 24 months. Measures the location and surface area of the pain.
Pain measurement 3 | Baseline, 4 months, 12months and 24 months
  Vas (visual analogue scale) 0, 4, 12, 24 months. Measures the pain in millimeters. 0 millimeters being no pain and 10 millimeters being the worst pain a patient can imagine.
Life quality: SRS-24 | Baseline, 4 months, 12months and 24 months
  SRS-24 scores (scoliosis research society's scoliosis patient questionnaire) at 0, 4, 12, and 24 months. The questionnaire was first developed to measure the life quality of scoliosis patients. The SRS-24 is a disease-specific HRQoL questionnaire used to assess the current state of the patient with scoliosis, and the effects of surgery, consisting of twenty-four questions, each with a grading of one to five points, with a maximum score of 120. The questionnaire evaluates seven domains: pain, general self-image, function from back condition, activity level, postoperative self-image, postoperative function and satisfaction.
Sit-up test | 4 months and 24 months
  Spinal mobility and strength tests will be done at 4months and 24 months follow-up visits. Sit-up test measures ab strength.The patient does as many sit-ups as he/she can. Maximum repetition will be 50 sit-ups.
back muscle test | 4 months and 24 months
  Spinal mobility and strength tests will be done at 4months and 24 months follow-up visits. In back muscle test patient will do back muscles and the measurement will be how many times one can do the movement. Maximum repetition will be 50.
squad test | 4 months and 24 months
  Spinal mobility and strength tests will be done at 4months and 24 months follow-up visits. In squad test it will be measured how many squads a patient can do. Maximum repetition will be 50 squads.
Back static hold | 4 months and 24 months
  Spinal mobility and strength tests will be done at 4months and 24 months follow-up visits. Patient will be in prone position and hold upper part of body up for as long as possible. It will be measured in seconds and the maximum hold up time is 240 seconds.
lumbar spine flexion | 4 months and 24 months
  Spinal mobility and strength tests will be done at 4months and 24 months follow-up visits. Lumbar spine flexion will be measured as patient bends forward in millimeters.
lumbar spine extension | 4 months and 24 months
  Spinal mobility and strength tests will be done at 4months and 24 months follow-up visits. Lumbar spine flexion will be measured as patient bends backward in millimeters.
lumbar spine rotation | 4 months and 24 months
  Spinal mobility and strength tests will be done at 4months and 24 months follow-up visits. Lumbar spine rotation will be measured with Myrins incliometer and the measurement will be grades and scaled between 0-360 degrees. The more rotation, the bigger the degree.
lumbar spine sidebend | 4 months and 24 months
  Spinal mobility and strength tests will be done at 4months and 24 months follow-up visits. Lumbar spine sidebending will be measured both sides in millimeters and the result is mediane of these.

CONTACTS AND LOCATIONS:
Overall Officials: Ella Virkki, Principal Investigator — pediatric surgeon
Locations (2):
- Finland (2):
  - Satakunta central hospital, Pori
  - Turku university hospital, Turku

IPD SHARING:
Plan to Share IPD: No